CLINICAL TRIAL: NCT01313728
Title: An Investigator-Blind, Phase 4 Study Assessing Mitigation of Facial Irritation When Comparing the Use of Two Acne Treatment Products (Retin-A Micro® 0.1 % Pump and Aczone®) With One Treatment Product (Retin-A Micro® 0.1 % Pump) Using a Split-Face Model
Brief Title: A Study That Evaluates the Decrease in Irritation When Using Additional Acne Treatment Products
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CA-P-7966
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
Keywords: Acne; Irritation
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone; Tretinoin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapsone plus Tretinoin Gel (Experimental): Dapsone gel, followed by tretinoin gel one hour later, applied once daily to the assigned side of the face for 2 weeks - all subjects participate in both arms in a split-face model
  Interventions: Drug: Dapsone plus Tretinoin Gel
- Tretinoin Gel Alone (Active Comparator): Tretinoin gel applied once daily to the assigned side of the face for 2 weeks - all subjects participate in both arms in a split-face model
  Interventions: Drug: Tretinoin Gel

INTERVENTIONS:
Drug: Dapsone plus Tretinoin Gel — Dapsone gel, followed by tretinoin gel one hour later, applied once daily to the assigned side of the face for 2 weeks
  Other Names: Aczone Gel 5% plus Retin-A Micro Gel 0.1% Pump
  Arms: Dapsone plus Tretinoin Gel
Drug: Tretinoin Gel — Tretinoin gel applied once daily to the assigned side of the face for 2 weeks
  Other Names: Retin-A Micro Gel 0.1% Pump
  Arms: Tretinoin Gel Alone

SUMMARY:
This study is to see if there's any difference in the amount of facial irritation when two acne products are used together on one side of the face, compared to one acne treatment product used alone on the other side of the face. All people participating in this trial will be required to return to the same study center every weekday for two weeks for the investigator to check for irritation on the face and to have the products applied - on weekends they will have to put them on at home. If one side of the face is more irritated than the other side, a picture will be taken as well.

DETAILED DESCRIPTION:
This is an investigator-blind, randomized, balanced study comparing two treatment regimens in a split-face model. All subjects will apply Retin-A Micro Gel (tretinoin) 0.1 % Pump, and Aczone Gel (dapsone) 5% daily to one side of the face (with 1 hour between applications, applying Aczone Gel first) and Retin-A Micro Gel 0.1 % Pump to the other side of the face in a randomized scheme for two consecutive weeks. Subjects will return to the study center daily for evaluation and for application of both products (weekend applications will be done at home). At each visit the subject will be evaluated and scored for irritation and cutaneous treatment effects. Subjects presenting with differences in irritation between one side of the face and the other will be photographed and have chromometer readings taken. A single treatment center is expected to enroll at least 24 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I, II or III with healthy skin as judged by the investigator
* Bilateral skin is clear of any confounding irritation, rashes, acne, rosacea, etc., prior to study start
* Subjects are willing to avoid applying emollients or cosmetics to the face 24 hours before they start, and during the study
* If subject is of childbearing potential, subject has been using a protocol-approved method of birth control for a certain amount of time, and is willing to continue using it throughout the study

Exclusion Criteria:

* Subjects who are pregnant or nursing, or intend to be during the study
* Subjects with any condition or medical history, or using any drug or medication, that might negatively affect the subject's safety or the validity of study results, either as listed in the protocol or in the opinion of the investigator
* Subjects who have facial hair that may obstruct or hinder the evaluation of any reactions
* Subjects who use any known photosensitizing agents

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lineberry, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Skin Study Center, Broomall, Pennsylvania, United States

REFERENCES:
- See also: FDA's Drug Finder — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: This was a single-group study with two treatment arms using a split-face model, i.e., all subjects received both interventions on opposite sides of the face.
Period: Informed Consent to Baseline
Arm/Group | Overall Study
Started | 26
Completed | 25 (One subject withdrew after signing informed consent, but prior to Baseline measurements being taken.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Baseline to Completion
Arm/Group | Overall Study
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex/Gender, Customized [Number; unit: Participants] — Gender was not a relevant measure for the trial, and was not recorded. Number reported reflects Participants in the overall study who were either Male or Female.
  Participants | 25
Region of Enrollment [Number; unit: participants]
  United States | 25
Fitzpatrick Score [Number; unit: Participants] — Skin type is categorized according to the Fitzpatrick skin type scale, which ranges from very fair (skin type I) to very dark (skin type VI). Only Skin Types I-III were included in this study.
  Participants
    Type I | 1
    Type II | 10
    Type III | 14

OUTCOME MEASURES:

1. Primary Outcome: Expert Grader Assessment - Erythema
Description: Ordinal erythema scores (on a scale of 0=none to 8=severe scaling and fissuring) were collected on weekdays for two weeks and the total daily score (for all subjects) was treated as a single interval measurement for comparative assessment between treatment regimens. Thus, for the total for the 25 Participants measured, minimum possible score reported below is 0 and maximum is 2000 (highest possible score of 8, times 10 days, times 25 subjects).
Time Frame: Baseline to 2 Weeks
Population: Intention to Treat (ITT)
Measure: Number; unit: Scores on a Scale
Groups:
- Dapsone Gel + Tretinoin Gel: Dapsone gel, followed by tretinoin gel one hour later, applied once daily to the assigned side of the face for 2 weeks - all subjects participate in both arms in a split-face model
- Tretinoin Gel Alone: Tretinoin gel applied once daily to the assigned side of the face
Arm/Group | Dapsone Gel + Tretinoin Gel | Tretinoin Gel Alone
Number analyzed (Participants) | 25 | 25
Scores on a Scale
  Day 0 = Baseline | 0.0 | 0.0
  Day 1 | 0.4 | 2.0
  Day 2 | 0.4 | 2.0
  Day 3 | 1.6 | 6.4
  Day 4 | 6.8 | 7.6
  Day 7 | 9.7 | 17.1
  Day 8 | 10.8 | 20.9
  Day 9 | 10.6 | 20.1
  Day 10 | 11.6 | 20.4
  Day 11 | 11.6 | 23.0
  Day 14 | 16.6 | 19.5

2. Primary Outcome: Expert Grader Assessment - Dryness
Description: Ordinal dryness scores (on a scale of 0=none to 8=deep) were collected on weekdays for two weeks and the total daily score (for all subjects) was treated as a single interval measurement for comparative assessment between treatment regimens. Thus, for the total for the 25 Participants measured, minimum possible score reported below is 0 and maximum is 2000 (highest possible score of 8, times 10 days, times 25 subjects).
Time Frame: Baseline to 2 Weeks
Population: Intention to Treat (ITT)
Measure: Number; unit: Scores on a Scale
Arm/Group | Dapsone Gel + Tretinoin Gel | Tretinoin Gel Alone
Number analyzed (Participants) | 25 | 25
Scores on a Scale
  Day 0 = Baseline | 0.0 | 0.0
  Day 1 | 0.6 | 1.8
  Day 2 | 1.7 | 2.5
  Day 3 | 3.5 | 8.1
  Day 4 | 12.6 | 14.2
  Day 7 | 14.8 | 19.9
  Day 8 | 18.5 | 25.6
  Day 9 | 13.6 | 23.0
  Day 10 | 20.4 | 37.6
  Day 11 | 17.3 | 37.6
  Day 14 | 23.5 | 28.3

3. Secondary Outcome: Subject Assessment - Burning/Stinging
Description: Ordinal burning/stinging scores (on a scale of 0=none to 3=severe) were collected on weekdays for two weeks and the total daily score (for all subjects) was treated as a single interval measurement for comparative assessment between treatment regimens. Thus, for the total for the 25 Participants measured, minimum possible score reported below is 0 and maximum is 750 (highest possible score of 3, times 10 days, times 25 subjects).
Time Frame: Baseline to 2 Weeks
Population: Intention to Treat (ITT)
Measure: Number; unit: Scores on a Scale
Arm/Group | Dapsone Gel + Tretinoin Gel | Tretinoin Gel Alone
Number analyzed (Participants) | 25 | 25
Scores on a Scale
  Day 0 = Baseline | 1.0 | 0.0
  Day 1 | 2.6 | 1.6
  Day 2 | 1.8 | 2.6
  Day 3 | 6.6 | 5.5
  Day 4 | 8.7 | 12.2
  Day 7 | 7.5 | 9.5
  Day 8 | 14.5 | 17.2
  Day 9 | 9.6 | 20.2
  Day 10 | 11.6 | 25.9
  Day 11 | 10.6 | 25.9
  Day 14 | 14.6 | 23.2

4. Secondary Outcome: Subject Assessment - Itching
Description: Ordinal itching scores (on a scale of 0=none to 3=severe) were collected on weekdays for two weeks and the total daily score (for all subjects) was treated as a single interval measurement for comparative assessment between treatment regimens. Thus, for the total for the 25 Participants measured, minimum possible score reported below is 0 and maximum is 750 (highest possible score of 3, times 10 days, times 25 subjects).
Time Frame: Baseline to 2 Weeks
Population: Intention to Treat (ITT)
Measure: Number; unit: Scores on a Scale
Arm/Group | Dapsone Gel + Tretinoin Gel | Tretinoin Gel Alone
Number analyzed (Participants) | 25 | 25
Scores on a Scale
  Day 0 = Baseline | 0.0 | 0.0
  Day 1 | 1.6 | 2.8
  Day 2 | 0.5 | 1.9
  Day 3 | 0.6 | 1.8
  Day 4 | 2.6 | 2.8
  Day 7 | 3.6 | 7.6
  Day 8 | 5.6 | 12.4
  Day 9 | 5.6 | 12.4
  Day 10 | 7.6 | 17.1
  Day 11 | 8.6 | 13.4
  Day 14 | 7.6 | 9.4

5. Secondary Outcome: Subject Assessment - Tightness
Description: Ordinal tightness scores (on a scale of 0=none to 3=severe) were collected on weekdays for two weeks and the total daily score (for all subjects) was treated as a single interval measurement for comparative assessment between treatment regimens. Thus, for the total for the 25 Participants measured, minimum possible score reported below is 0 and maximum is 750 (highest possible score of 3, times 10 days, times 25 subjects).
Time Frame: Baseline to 2 Weeks
Population: Intention to Treat (ITT)
Measure: Number; unit: Scores on a Scale
Arm/Group | Dapsone Gel + Tretinoin Gel | Tretinoin Gel Alone
Number analyzed (Participants) | 25 | 25
Scores on a Scale
  Day 0 = Baseline | 0.0 | 0.0
  Day 1 | 1.5 | 1.8
  Day 2 | 1.5 | 2.9
  Day 3 | 2.6 | 4.7
  Day 4 | 5.7 | 8.5
  Day 7 | 8.6 | 12.5
  Day 8 | 12.5 | 19.0
  Day 9 | 11.6 | 17.2
  Day 10 | 12.5 | 20.0
  Day 11 | 9.6 | 15.3
  Day 14 | 10.5 | 14.4

6. Secondary Outcome: Facial Tolerance
Description: All interval measurements were combined for comparative assessment between treatment regimens. Facial tolerance is the sum of scores from Erythema, Dryness, Burning/Stinging, Itching, and Tightness assessments, reported in Outcome Measures 1-5. Thus, for the total for the 25 Participants measured, minimum possible score reported below is 0 and maximum is 6250 (highest possible combined score of 25, times 10 days, times 25 subjects).
Time Frame: Baseline to 2 Weeks
Measure: Number; unit: Scores on a Scale
Arm/Group | Dapsone Gel + Tretinoin Gel | Tretinoin Gel Alone
Number analyzed (Participants) | 25 | 25
Scores on a Scale
  Day 0 = Baseline | 1.0 | 0.0
  Day 1 | 6.7 | 10.0
  Day 2 | 5.9 | 11.9
  Day 3 | 14.9 | 26.5
  Day 4 | 36.4 | 45.3
  Day 7 | 44.2 | 66.6
  Day 8 | 61.9 | 95.1
  Day 9 | 51.0 | 93.9
  Day 10 | 63.7 | 124.6
  Day 11 | 57.7 | 115.2
  Day 14 | 72.8 | 94.8

ADVERSE EVENTS:
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=25)
Irritation (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days